CLINICAL TRIAL: NCT05286567
Title: An Investigator Initiated, Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Proof-Of-Concept Study to Assess the Safety and Efficacy of a Novel HSP90 Inhibitor (RGRN-305) in the Treatment of Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Double-blind Placebo-controlled Randomized Trial Evaluating the Efficacy and Safety of a Novel HSP90 Inhibitor (RGRN-305) in the Treatment of Moderate to Severe Hidradenitis Supppurativa.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Hakim Ben Abdallah, M.D., Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGRN-305-002; 2021-000881-13 (EudraCT Number)
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGRN-305 (Experimental): 1 tablet of 250mg RGRN-305 once daily for 16 weeks
  Interventions: Drug: RGRN-305
- Placebo (Placebo Comparator): 1 tablet of placebo once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGRN-305 — Heat shock protein 90 inhibitor
  Arms: RGRN-305
Drug: Placebo — Placebo (blinded)
  Arms: Placebo

SUMMARY:
This is a 16-week treatment, randomized, double-blind, proof-of-concept study designed to assess the safety and efficacy of RGRN-305 compared to placebo for use in future efficacy Phase 2 trials.

Male or female subjects aged 18 years or older with moderate to severe hidradenitis suppurativa will be included in this study.

Objectives are to determine the efficacy and safety of RGRN-305 in patients with moderate to severe hidradenitis supppurativa.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to be enrolled in the study if they meet all of the following criteria at the Screening and Baseline (Day 0) Visits, unless specified otherwise:

1. Men or women aged 18 years or older at the time of consent.
2. Subject has a history of onset of hidradenitis suppurativa for at least 6 months prior to Baseline (Day 0) Visit.
3. Subject has hidradenitis suppurativa with at least 5 inflammatory nodules or abscesses (total AN count) in at least 2 distinct anatomic areas, both at Screening and Baseline (Day 0) Visits. Furthermore, one additional inflammatory nodule must be present for collection of skin biopsies.
4. Subjects (women and men) involved in any sexual intercourse that could lead to pregnancy must agree to use an effective contraceptive method from at least 4 weeks before Baseline (Day 0) until at least 4 weeks after the last study product administration for the duration of the study. Effective contraceptive methods are: systemic hormonal contraceptives (oral contraceptive, patch, vaginal ring, injectables, or implants), intrauterine devices, vasectomy, or barrier methods of contraception in conjunction with spermicide. Hormonal contraceptives must be on a stable dose for at least 4 weeks before Baseline (Day 0).

   Note: Woman of non-childbearing potential are as follows:
   * Women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation).
   * Women ≥ 60 years of age.
   * Women > 40 and < 60 years of age who have had a cessation of menses for at least 12 months and a follicle-stimulating hormone (FSH) test confirming non-childbearing potential (FSH ≥ 40 mIU/mL) or cessation of menses for at least 24 months without FSH levels confirmed.

   Protocol RGRN-305 - Safety and Efficacy of RGRN-305 in HS Page 13 of 61 Protocol version 3.2: 13 September 2021
5. Women of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at Baseline (Day 0).
6. Subject must have negative tuberculosis (TB) infection tests. Subjects will be evaluated for latent TB infection with a purified protein derivative (PPD) test, T-spot test or a Quantiferon Gold test, and with a chest x-ray, if one has not been performed in the last 6 months. Subject who demonstrates evidence of latent TB infection (either PPD ≥ 5 mm of induration or positive Quantiferon Gold or T-spot test, irrespective of Bacillus Calmette-Guérin (BCG) vaccination status and negative chest x-rays findings for active TB, or suspicious chest x-ray findings) will not be allowed to participate in the study.
7. Subject must be willing to participate and must be capable of giving informed consent, and the consent must be obtained prior to any study-related procedures.

Exclusion Criteria:

1. Female subject who is breastfeeding, pregnant, or who is planning a pregnancy during the study.
2. Subject has a history of skin disease or presence of a skin condition that, in the opinion of the investigator, would interfere with the study assessments.
3. Subject is known to have immune deficiency or is immunocompromised.
4. Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Baseline (Day 0). Subjects with successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
5. Subject has had a major surgery within 8 weeks prior to Baseline (Day 0) or has a major surgery planned during the study.
6. Subject has any clinically significant medical condition including ongoing infections, or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
7. Subject has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values ≥ 2 times the upper limit of normal (ULN) at Screening.
8. Subject has absolute neutrophil count ≤ 1.5 X 109/L or platelet count ≤ 100 X 109/L at Screening.
9. Subject has a history of clinically significant anemia or hemoglobin (Hgb) value ≤ 10 g/dL (6.21 mmol/dL) at Screening.
10. Subject has a creatine clearance ≤ 60 mL/min at Screening (calculated with Cockcroft-Gault formula).
11. Subject with positive results for hepatitis B surface antigens (HBsAg), anti-hepatitis B core antibodies (anti-HBc), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
12. Subject has a known or suspected allergy to RGRN-305 or any component of the investigational product.
13. Subject has a history of clinically significant drug or alcohol abuse in the last year prior to Baseline (Day 0) Visit.
14. Subject is currently receiving an investigational product or device or has received one within 4 weeks prior to Baseline (Day 0) Visit.
15. Subject has received a live attenuated vaccine within 4 weeks prior to Baseline (Day 0) Visit or plan to receive a live attenuated vaccine during the study and up to 1 month after the last study drug administration.
16. Subject has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
17. Subject has a history of hypertrophic scarring or keloid formation in scars or suture sites.
18. Known inability or unavailability of a subject to complete required study visits during study participation.
19. A psychiatric condition (e.g., suicidal ideation), chronic alcohol, or drug abuse problem, determined from the subject's medical history, which, in the opinion of the investigator, may pose a threat to subject compliance.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR-50) score | Week 16

SECONDARY OUTCOMES:
Percentage of subjects with Hidradenitis Suppurativa Physician's Global Assessment (HS-PGA) scores of clear or minimal | Week 2, 4, 8, 12, 14, 16, and 20.
Percentage of subjects achieving HiSCR-50, HiSCR-75, and HiSCR-90 | Week 2, 4, 8, 12, 14, 16, and 20.
Changes from Baseline in the Dermatology Life Quality Index (DLQI) total score | Week 4, 8, 12, 16, and 20.
  Minimum score: 0 (no effect at all on patient's life) Maximum score: 30 (extremely large effect on patient's life)
Changes from Baseline in the Pain Numerical Ranging score | Weeks 4, 8, 12, 16, and 20
  Minimum score: 0 (No pain) Maximum score: 10 (worst pain)
Change and percent change from Baseline in lesion counts (abscess count, inflammatory nodule count, AN count, and draining tunnel count). | Week 2, 4, 8, 12, 14, 16, and 20.
Change from Baseline in skin biomarkers | Week 16.
Change from Baseline in blood biomarkers | Week 4, 8, 12, and 16.
Incidence of treatment-emergent adverse events (TEAEs). | Week 20
Incidence of related TEAEs. | Week 20

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ben Abdallah H, Bregnhoj A, Emmanuel T, Ghatnekar G, Johansen C, Iversen L. Efficacy and Safety of the Heat Shock Protein 90 Inhibitor RGRN-305 in Hidradenitis Suppurativa: A Parallel-Design Double-Blind Trial. JAMA Dermatol. 2024 Jan 1;160(1):63-70. doi: 10.1001/jamadermatol.2023.4800. PMID 38055242